CLINICAL TRIAL: NCT05326269
Title: Acute Tocolysis With Terbutaline vs Placebo Prior to Emergency Caesarean Delivery for Suspected Intrauterine Fetal Compromise
Brief Title: Acute Tocolysis With Terbutaline for Suspected Fetal Distress
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Kemaman (Other)
Responsible Party: Principal Investigator, Zahar Azuar Zakaria, Principal investigator, Consultant Obstetrician, Hospital Kemaman
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NMRR-16-1985-331
Record Dates: First submitted 2022-03-22; First posted 2022-04-13 (Actual); Last update posted 2022-04-13 (Actual); Status verified 2022-04

CONDITIONS: Nonreassuring Fetal Status
Keywords: fetal resuscitation; acute tocolysis; fetal distress; cesarean section
MeSH Terms: conditions — Fetal Distress | interventions — Terbutaline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: The participants are randomly assigned a number (generated using an online random number generator) and given an opaque envelope containing instructions for study drug or placebo administration. The envelope will be opened by a nurse who prepared the injection in a treatment room, separated from the Labour Suite. The doctors managing the cases, the surgeons who performed the surgeries, the anaesthetists and the patients themselves were blinded against the injection given
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Active Comparator): Terbutaline 0.5 mls (0.25 mg) , subcutaneously
  Interventions: Drug: Terbutaline
- Control group (Placebo Comparator): Placebo (normal saline) 0.5 mls , subcutaneously
  Interventions: Drug: Terbutaline

INTERVENTIONS:
Drug: Terbutaline — Subcutaneous injection
  Other Names: beta mimetic

SUMMARY:
The trial was to determine the effect of administrating subcutaneous terbutaline prior to emergency caesarean delivery for suspected fetal distress

DETAILED DESCRIPTION:
The trial was a double-blinded, placebo-controlled study using subcutaneous terbutaline for acute tocolysis prior to emergency caesarean delivery in suspected fetal distress. The intervention (subcutaneous terbutaline) was compared to placebo looking at the neonatal and maternal outcomes.

The primary outcome was the proportion of babies with neonatal acidosis (based on umbilical artery blood sampling at delivery). Other outcome of interest were the mean cord pH and base excess, the Apgar score at 5 minutes after delivery, he proportion of babies requiring intubation and admission to the Neonatal Intensive Care Unit. The maternal outcomes of interest were the changes in mean arterial pressure (before and after the drug or placebo injection), the maternal heart rate changes, the estimated blood loss, and the hematocrit changes.

ELIGIBILITY:
Inclusion Criteria:

* term singleton pregnancy
* cephalic presentation
* in labour with cervix dilatation > 4cm and regular uterine contractions of 3 or more 10 min
* abnormal fetal heart rate status diagnosed using standard electronic FHR according to NICE guideline (2014)
* acceptance of participation by the signing of a written consent.

Exclusion Criteria

* maternal cardiopathy
* hyperthyroidism
* abruptio placentae or other placental accidents
* hypertensive disease of pregnancy
* hyperstimulation with oxytocin
* multiple gestation
* abnormal fetus planned for conservative management
* evidence of intrauterine growth restriction
* patient on medication which will interact with terbutaline (tricyclic antidepressants, beta-blockers, diuretics and sympathomimetic medicine).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2017-04-23 (Actual); Primary Completion 2019-09-15 (Actual); Study Completion 2019-09-15 (Actual)

PRIMARY OUTCOMES:
Neonatal acidosis | within 1 hour of delivery
  Umbilical artery acidosis

SECONDARY OUTCOMES:
Neonatal acid base status | within 1 hour of delivery
  Mean umbilical artery pH & base excess
Neonatal Apgar score | 5 minutes after delivery
  Mean Apgar score at 5 minutes of life
Neonatal intensive care unit admission | Within 24 hours of delivery
  Number of babies admitted to neonatal intensive care unit
Maternal blood pressure | Within 1 hours after drug administration
  Mean maternal arterial pressure (before and after drug or placebo administration)
Maternal heart rate | Within 1 hours after drug administration
  Mean maternal heart rate changes (before and after drug or placebo administration)
Blood loss | Within 24 hours of delivery
  Mean estimated blood loss
Hematocrit change | Within 24 hours of delivery
  Mean hematocrit changes before and after cesarean section

CONTACTS AND LOCATIONS:
Overall Officials: Zahar A Zakaria, MD, Principal Investigator — Hospital Kemaman
Locations (1):
- Hospital Kemaman, Kuala Terengganu, Terengganu, Malaysia

IPD SHARING:
Plan to Share IPD: No
Upon request

REFERENCES:
- [Background] Patriarco MS, Viechnicki BM, Hutchinson TA, Klasko SK, Yeh SY. A study on intrauterine fetal resuscitation with terbutaline. Am J Obstet Gynecol. 1987 Aug;157(2):384-7. doi: 10.1016/s0002-9378(87)80178-3. PMID 3303936
- [Background] Ingemarsson I, Arulkumaran S, Ratnam SS. Single injection of terbutaline in term labor. I. Effect on fetal pH in cases with prolonged bradycardia. Am J Obstet Gynecol. 1985 Dec 15;153(8):859-65. doi: 10.1016/0002-9378(85)90690-8. PMID 4073156
- [Background] Leathersich SJ, Vogel JP, Tran TS, Hofmeyr GJ. Acute tocolysis for uterine tachysystole or suspected fetal distress. Cochrane Database Syst Rev. 2018 Jul 4;7(7):CD009770. doi: 10.1002/14651858.CD009770.pub2. PMID 29971813
- [Background] Pullen KM, Riley ET, Waller SA, Taylor L, Caughey AB, Druzin ML, El-Sayed YY. Randomized comparison of intravenous terbutaline vs nitroglycerin for acute intrapartum fetal resuscitation. Am J Obstet Gynecol. 2007 Oct;197(4):414.e1-6. doi: 10.1016/j.ajog.2007.06.063. PMID 17904983
- [Result] Buckley VA, Wu J, De Vries B. Outcomes following acute tocolysis prior to emergency caesarean section. Aust N Z J Obstet Gynaecol. 2020 Dec;60(6):884-889. doi: 10.1111/ajo.13170. Epub 2020 May 6. PMID 32378185
- [Result] Magann EF, Cleveland RS, Dockery JR, Chauhan SP, Martin JN Jr, Morrison JC. Acute tocolysis for fetal distress: terbutaline versus magnesium sulphate. Aust N Z J Obstet Gynaecol. 1993 Nov;33(4):362-4. doi: 10.1111/j.1479-828x.1993.tb02109.x. PMID 8179541